CLINICAL TRIAL: NCT04663997
Title: A Randomized Phase II Study of 177 LuPSMA-617 vs Docetaxel in Patients With Metastatic Castration-Resistant Prostate Cancer and PSMA-Positive Disease
Brief Title: 177 LuPSMA-617 vs Docetaxel in Metastatic Castration Resistant and PSMA-Positive Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Prostate Cancer Canada (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR21
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-10

CONDITIONS: Prostate Cancer
Keywords: mCRPC; docetaxel; 177Lu-PSMA-617; radioligand therapy; metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 177 Lu-PSMA-617 (Experimental)
  Interventions: Drug: 177Lu-PSMA-617
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — IA of 7.4GBq (± 10%) IV every 6 weeks; maximum 6 cycles
  Arms: 177 Lu-PSMA-617
Drug: Docetaxel — 75mg/m2 IV every 3 weeks maximum 12 cycles
  Arms: Docetaxel

SUMMARY:
177Lu PSMA 617 is a new type of therapy which is designed to deliver high doses of radiation directly to prostate cancer sites in the body. The purpose of this study is to find out whether 177Lu PSMA 617can slow the growth of prostate cancer compared to standard chemotherapy treatment

DETAILED DESCRIPTION:
The standard or usual treatment for this disease is a chemotherapy drug called docetaxel, given by intravenous every 3 weeks, for up to 12 treatments.

177Lu-PSMA-617 is a new type of therapy for prostate cancer. Laboratory tests show that it may help slow the growth of prostate cancer. 177Lu-PSMA-617 has been shown to shrink tumours in animals and has been studied in limited numbers of men with prostate cancer and seems promising but it is not clear if it can offer better control of prostate cancer compared to docetaxel chemotherapy .

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of prostate cancer with no evidence of small cell component
* Patients must have castration resistance and metastatic disease with evidence of biochemical or imaging progression in the setting of surgical/medical castration
* Progression on treatment with abiraterone and/or enzalutamide, or similar next-generation androgen receptor (AR) targeted therapy
* Evidence of PSMA positive metastatic disease, as assessed on PSMA-PET imaging studies obtained as part of other clinical trial protocols are mandated, provided they are obtained within a timeframe that meets the requirements of this study. The radiopharmaceuticals must be based on a lysine-urea-glutamate backbone, with a 18F or 68Ga radionuclide label.
* Prior orchiectomy, or if on LHRH agonist/antagonist then testosterone < 1.7 nmol/L
* Adequate organ function
* Recover from all previous cancer treatment toxicities to grade ≤ 2 (as per CTCAE v5.0)
* Male subject ≥ 18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria:

* Prior treatment with chemotherapy for castration-resistant disease or prior chemotherapy in the castration-sensitive (hormone-sensitive) setting ≤ 1 year prior to enrollment.
* Prior treatment with 177Lu-PSMA (including other radiolabeled therapeutic PSMA-ligands) or radio-immunotherapy. Prior treatment with radium-223 is allowed but requires a minimum of a 6-month interval between the last dose of radium-223 and enrollment.
* Radiotherapy to target lesions (measurable disease) ≤ 12 weeks prior to enrolment.
* Presence of majority (> 50% of extra-osseous lesions) or large (> 5 cm) soft tissue lesions that are negative on PSMA-Ligand PET/CT or PSMA-Ligand PET/MR
* Known parenchymal brain metastases
* Active epidural disease (treated epidural disease is permitted)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Clinically significant cardiac disease
* Major surgery within 4 weeks of starting study treatment
* Patients with a history of hypersensitivity to the study drug or components
* Patients with a clinically significant medical condition which, in the opinion of the treating physician, makes it undesirable for the patient to participate in the study or which could jeopardize compliance with study requirements including, but not limited to: ongoing or active infection, significant uncontrolled hypertension, or sever psychiatric illness/social situations.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2025-08-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 3 years

SECONDARY OUTCOMES:
Progression-free survival rate at 6 months defined by PSA | 6 months
Progression-free survival rate at 6 months defined by PCWG 3 | 6 months
Progression-free survival rate at 6 months defined by RECIST 1.1 | 6 months
Second rPFS in patients who meet the criteria for rPFS and cross over to the alternate therapy | 3 years
Time to commencement of third line therapy | 3 years
Overall Survival | 3 years
Proportions of patients with decreased PSA from baseline and the magnitude of change | 3 years
  e.g. ≥ 30%, ≥ 50%, ≥ 90% decline from baseline
Clinical benefit rate (CBR) > 24 weeks (RECIST v1.1). | 3 years
Response duration including partial response, complete response or stable disease > 24 (RECIST v1.1) | 3 years
Adverse event (AE) profile (CTCAE v5.0) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada; Francois Benard, Study Chair — BCCA - Vancouver Cancer Centre, BC Canada; Fred Saad, Study Chair — CHUM-Centre Hospitalier de l'Universite de Montreal, Canada
Locations (10):
- Canada (10):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Program, London, Ontario
  - Odette Cancer Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - The Jewish General Hospital, Montreal, Quebec
  - Hotel-Dieu de Quebec, Québec, Quebec
  - CIUSSS de l'Estrie - Centre hospitalier, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No
Subject to CCTG Policy